CLINICAL TRIAL: NCT04910906
Title: Prospective Post-market Clinical Follow up Study to Assess Efficacy and Safety of Ectoin® Vaginal Gel (EIC01) for Symptomatic Treatment of Vaginal Atrophy in Post-menopausal Women
Brief Title: Non-Interventional Multicentre Post-market Study of Ectoin® Vaginal Gel for Symptomatic Treatment of Vaginal Atrophy
Acronym: EIC01-PMCF
Status: Completed | Type: Observational
Sponsor: Bitop AG (Industry)
Responsible Party: Sponsor
Other Study IDs: btph-045-2020-EIC01
Record Dates: First submitted 2021-05-25; First posted 2021-06-02 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Vaginal Atrophy
Keywords: vaginal atrophy; vaginal dryness; post-menopausal symptoms; post-menopausal Vaginal health

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ectoin® Vaginal Gel — Ectoin® Vaginal Gel is a clear, non-hormonal moisturizing gel containing only active ingredient Ectoin® for the relief of vaginal dryness/vaginal atrophy.
  Other excipients in the formulation include:
  Hydroxyethylcellulose (Gelling agent) Lactic acid (90 %) (pH stabiliser) DL-Sodium lactate (Buffer substance) Sodium benzoate (preservative) Propylene glycol (Humectant)

SUMMARY:
The goal of this multi-centre, prospective, open label, single arm, observational post-market clinical follow-up study (§23b of the MPG (German Medical Act) MDD 93/42/EEC and ISO14155:2020) is to investigate and evaluate the clinical efficacy of Ectoin® Vaginal gel (EIC01) to retain/restore the natural moisturization in the vaginal lumen and to alleviate vaginal atrophy symptoms.

DETAILED DESCRIPTION:
A multi-centre, prospective, open label, single arm, observational post-market clinical follow-up study according to §23b of the MPG (German Medical Act) and conforming to MDD 93/42/EEC and ISO14155:2020.

Study participation will be offered to patients with symptoms of vaginal atrophy for which Ectoin® Vaginal Gel is indicated. Screening period might take up to 14 days. If the patient, at the screening visit, complies with all the inclusion criteria (except inclusion criterion No. 4 which is to be confirmed at the Baseline Visit) and she has signed the informed consent, she will be enrolled, and baseline visit will be performed on the same day.

The Ectoin® Vaginal Gel will be used for 20 days and in accordance with the IFU . Visits are scheduled on day 1, 5, and 20, at which the treatment is ended (End of treatment - EoT). Follow-up (FU) visit is planned on Day 23. Patient will record her symptoms and number of applied doses in the patient diary on daily basis, preferably around a specific time which has to be followed throughout the entire study period. Overall, participation will take at least 23 (+2) days and 37 (+2) days at maximum. The enrolment period will take 2 months. The total duration of the study is expected to be approximately 3-6 months.

The efficacy and safety of Ectoin® Vaginal Gel (EIC01) in the alleviation of vaginal atrophy symptoms will be evaluated in this study. Efficacy will be evaluated based on the improvement of Vaginal Atrophy symptoms at post-treatment measurements as compared to baseline values.

Primary endpoint is to evaluate the efficacy of the EIC01 product by analysing the difference in the sum scores of Vaginal Health Index (VHI) indicating both subjective and objective improvement in the vaginal atrophy condition after multiple application.

Secondary Endpoint:

* Improvement in individual and sum score of VAS for vaginal atrophy symptoms (feeling of dryness, itching, burning, pain during sexual intercourse) after single (immediate effect) and multiple applications
* Assessment of vaginal atrophy impact on life through Q/A
* Assessment of product acceptance and overall satisfaction through Q/A (on 20 day - V2) • Long-term treatment effect based on rate of improvement compared to baseline condition determined by subjective and objective assessments (5 days, 20 days and 23 days).
* Long-lasting effect assessed during follow-up by subjective and objective assessments on day 23.
* The treatment safety will be assessed by observation and documentation of adverse events and device deficiencies.
* Local tolerability will be assessed both by physician and patient using five-point scale (excellent, good, moderate, poor, bad).

ELIGIBILITY:
Inclusion Criteria:

* Menopausal women 50 years of age or older with no menstruation for at least 12 months.
* Self-reported vaginal atrophy symptoms and presence of all 4 common vaginal atrophy symptoms i.e., feeling of vaginal dryness, itching, burning sensation and dyspareunia.
* Sexually active women.
* Vaginal atrophy clinically confirmed through physical examination of vagina and vaginal pH; pH ≥ 5 and VHI ≤ 15.
* Patient who qualifies for Ectoin® Vaginal Gel treatment according to the approved indication and in physician's opinion the participant will benefit from this treatment.
* Signed informed consent.
* Willingness of the participants to actively participate in the study and to come to the scheduled visits.
* Willingness of the participants to continue the application of EIC01 in the test area throughout the course of the study and to avoid forbidden treatment.

Exclusion Criteria:

* Women reporting systemic post-menopausal symptoms (eg. hot flushes, sleep disturbances, slowed metabolism etc.) in addition to clinically confirmed vaginal atrophy.
* Women who had not performed a cervical cytology in the last year to rule out underlying critical condition.
* Vaginal infections (in past 8 weeks)
* Women taking systemic hormone replacement or pills within last 6 months.
* Patients with concomitant clinically important medical disease according to the investigator's opinion that might interfere with patient safety or evaluation of study results; that includes but not limited to endometrial hyperplasia or cancer; undiagnosed vaginal bleeding; liver or kidney disorder; thromboembolic disorders; cerebrovascular accident, stroke, or transient ischemic attack; myocardial infarction or ischemic heart disease; malignancy; endocrine disease or any clinically important abnormalities on (if any) screening physical examination, mammogram, electrocardiogram (ECG), or laboratory tests (indicative of any vaginal infection).
* Participation in any other clinical study within the last 4 weeks prior to the baseline visit.
* Previous incident or knowledge of possible hypersensitivity or allergic reactions to any of the components of EIC01.
* Previous treatment with other local non-hormonal moisturisers/hormonal products within 1 month or use of lubricants within 1 week prior to inclusion.
* Treatment with systemic medications for other non-related health condition which might impact the study results e.g. glucocorticosteroids, antibiotics etc. which has the potential to bring about change in vaginal environment.
* Medical or mental condition for which in the opinion of the physician, patient will not be able to fulfil questionnaires independently or to adhere to instructions and procedures in accordance with the study protocol

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: post-menopausal women of 50 years or above with no menstruation > 12 months and self-reporting/complaining of vaginal atrophy symptoms.
  Vaginal atrophy (VA) is a condition occurring due to the deteriorating structural and functional integrity of the vulvovaginal epithelium. It is commonly observed in menopausal and post-menopausal women and associated with an increased feeling of vaginal dryness and frequent/persistent irritation (burning sensation and pruritus) and pain on penetration (dyspareunia) in the vagina. VA also results in cytomorphological changes of the vaginal mucosa; however, it is the vulvovaginal symptoms associated with VA which are considered most bothersome, such as dryness, itching, burning sensation, and dyspareunia (pain during sexual penetration).
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2022-02-09 (Actual); Study Completion 2022-02-09 (Actual)

PRIMARY OUTCOMES:
Change in Vaginal Health Index (VHI) Score | treatment 20 days + FU 3 to 5 days
  Assessment of vaginal lumen condition by gynaecologist from baseline to end of study on 20th day of application and thereafter, follow-up assessment in 3-5 days from end of treatment. The VHI components are graded from 1-5; where 1 indicating worst possible and 5 indicating best possible conditions.

SECONDARY OUTCOMES:
Change in vaginal pH | 20+ (3-5) days FU
  Descriptive account of the vaginal pH as determined by the investigator during the visits using pH indicator strips of range 4.0 -7.0 pH
Change in severity of VA symptoms (vaginal irritation, itching, vaginal dryness, and dyspareunia) | 20+ (3-5) days FU
  Patient reported outcome on a VAS scare graded from 0-10; 0 = no problem and 10 = extremely unbearable
Change in total score in Quality of Life evaluation parameters | 20+ (3-5) days FU
  MCQ (multiple choice questions) format to choose the answer that corresponds best to the patient's situation. Patient have to choose between 4 options defining varying state possible outcome relevant to each specific question.
Change in score of overall vaginal atrophy condition | 20+ (3-5) days FU
  Patient reported outcome on a VAS scare graded from 0-10; 0 = no problem and 10= extremely unbearable
Change in score of symptoms based rating on need for treatment | 20+ (3-5) days FU
  Patient reported outcome on a VAS scare graded from 0-10; 0 = no at all and 10 = extreme need
Overall tolerability assessments | 20 days
  tolerability assessments (investigator and/or patient) on a 5-point scale;
  1 = excellent (no reaction), 2 = good (small reaction that spontaneously resolves), 3 = moderate (reaction tolerated with difficulty by the subject), 4 = poor (reaction needing interruption of treatment), 5 = bad (serious reaction)
Number of AEs and assessment of intensity, causality and seriousness of Adverse Events | 20 days
  The adverse events will be classified as non-serious adverse event or serious adverse event (SAE), the intensity will be graded as mild, moderate, severe, life threatening or fatal. The causality will be classified as definitely, probably, possibly, or not related and in case of none of the above should be defined as an unknown relationship.

CONTACTS AND LOCATIONS:
Overall Officials: Shatadal Sen, MSc., Study Chair — Project Manager (Medical Device Development)
Locations (1):
- bitop AG, Dortmund, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided